CLINICAL TRIAL: NCT02149420
Title: A Single Dose, Double-blind, Placebo-controlled, Parallel Study to Assess the Pharmacodynamics, Pharmacokinetics and Safety and Tolerability of VAY736 in Patients With Primary Sjögren's Syndrome
Brief Title: PD of VAY736 in Patients With Primary Sjögren's Syndrome
Acronym: CVAY736X2201
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVAY736X2201; 2013-000250-22 (EudraCT Number)
Record Dates: First submitted 2013-09-09; First posted 2014-05-29 (Estimated); Results first posted 2019-02-12 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Primary Sjögren's Syndrome
Keywords: primary Sjögren's syndrome, pharmacodynamics
MeSH Terms: interventions — ianalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment was unblinded at an individual patient level at Week 24 to determine their progress in the study (follow-up, open-label VAY736 or End of Study Visit).
Oversight: Data Monitoring Committee: No

ARMS (3):
- VAY736 3 mg/kg (Experimental): single dose iv of VAY736 at a dose of 3mg/kg
  Interventions: Drug: VAY736
- VAY736 10 mg/kg (Experimental): single dose iv of VAY736 at a dose of 10mg/kg
  Interventions: Drug: VAY736
- Placebo (Placebo Comparator): single dose iv of Placebo. At Week 24 patients were offered to receive open label VAY736 10 mg/kg.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VAY736
  Arms: VAY736 10 mg/kg; VAY736 3 mg/kg
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study was designed to evaluate the safety, tolerability, pharmacokinetics and therapeutic efficacy of a single intravenous infusion of VAY7346 monoclonal antibody in pSS patients

DETAILED DESCRIPTION:
Patients were enrolled in 2 sequential cohorts:

Cohort 1: 6 patients received 3 mg/kg or Placebo (2:1 ratio) Cohort 2: 21 patients received 10 mg/kg, 3 mg/kg or Placebo (6:1:3 ratio)

At week 24 the blind was broken to assess continuation in the trial:

* If a patient received VAY736 and their B cell recovery was demonstrated at Week 24, then patients completed the trial.
* If a patient received VAY736 and their B cell recovery was NOT demonstrated at Week 24, then patients were followed up until B cell recovery was demonstrated
* If a patient received placebo, they were offered the option of receiving open-label VAY736 (10 mg/kg) in a separate treatment arm.

ELIGIBILITY:
INCLUSION CRITERIA:

* Fulfilled revised European US consensus criteria for pSS
* ESSDAI value ≥ 6
* Elevated serum titers at screening of ANA (≥ 1:160)
* Seropositive at screening for anti-SSA and/or anti-SSB antibodies
* Stimulated whole salivary flow rate at screening of > 0 mL/min

EXCLUSION CRITERIA:

- Prior or previous use of (specific dosages and intervals prior to study start may apply): B-cell depleting therapy (e.g., rituximab), Prednisone, anti-BAFF mAb, CTLA4-Fc Ig (abatacept), anti-TNF-α mAb, cyclophosphamide, azathioprine and medications known to cause dry mouth.

Hydroxychloroquine or methotrexate in a consistent dose for ≥ 3 months prior to randomization is allowed

* Active or recent history of clinically significant infection
* Vaccination within 2 month prior to study
* History of primary or secondary immunodeficiency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-05-23 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Berlin, Germany

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=419

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 27 patients were enrolled and randomized into the study at one site in Germany.
Pre-assignment Details: The patients were enrolled in 2 sequential cohorts:
  Cohort 1: Six patients were randomized to receive a single dose iv of VAY736 at a dose of 3mg/kg or placebo at a 2:1 ratio.
  Cohort 2: Twenty one patients were randomized to receive a single iv dose of VAY736 at a dose of 10.0 mg/kg or 3.0 mg/kg or placebo at a 6:1:3 ratio.
Groups:
- Placebo: single dose iv of Placebo (+ Option to receive Open label VAY736 10 mg/kg at Week 24)
Period: Core Study
Arm/Group | Placebo | VAY736 3 mg/kg | VAY736 10 mg/kg
Started | 9 | 6 | 12
Safety Analysis Set (all patients that received study drug) | 9 | 6 | 12
PK Analysis Set (at least one valid PK concentration measurement) | 5 (for patients entering open label VAY736 10 mg/kg at Week 24) | 6 | 12
PD (Pharmacodynamics) Analysis Set (all patients with PD data, who received at least one dose of study drug.) | 9 | 6 | 12
Completed | 9 | 5 | 10
Not Completed | 0 | 1 | 2
Not completed — Administrative problems | 0 | 1 | 2
Period: Open Label VAY736 10 mg/kg Extension
Arm/Group | Placebo | VAY736 3 mg/kg | VAY736 10 mg/kg
Started | 5 (Patients received single dose of VAY736 10mg/kg at Week 24.) | 0 (Only patients origianally randomized to Placebo were allowed to enter this Period.) | 0 (Only patients origianally randomized to Placebo were allowed to enter this Period.)
Completed | 4 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Administrative problems | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: single dose iv of Placebo
- Total: Total of all reporting groups
Arm/Group | Placebo | VAY736 3 mg/kg | VAY736 10 mg/kg | Total
Number analyzed (Participants) | 9 | 6 | 12 | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.7 (11.29) | 46.8 (8.75) | 55.3 (13.35) | 50.5 (12.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 11 | 23
  Male | 2 | 1 | 1 | 4
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 9 | 6 | 12 | 27

OUTCOME MEASURES:

1. Primary Outcome: Change in EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI)
Description: The effect of VAY736 on clinical disease activity was measured by the change in ESSDAI (EULAR Sjögren's syndrome disease activity index) between baseline and week 12. The instrument contains 12 organ-specific domains contributing to disease activity. For each domain, features of disease activity are scored in 3 or 4 levels according to their severity. These scores are then summed across the 12 domains in a weighted manner to provide the total score (range 0-123). A reduction from baseline indicates improvement in patients.
Time Frame: Baseline, week 12
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- VAY736 Combined: Combining VAY736 3mg/kg and VAY736 10mg/kg
Arm/Group | Placebo | VAY736 3 mg/kg | VAY736 10 mg/kg | VAY736 Combined
Number analyzed (Participants) | 9 | 6 | 12 | 18
units on a scale
  Baseline | 11.1 (4.08) | 14.5 (9.44) | 11.5 (4.38) | 12.5 (6.38)
  Week 12 | 10.2 (5.29) | 10.7 (7.69) | 10.0 (5.36) | 10.2 (6.01)
  Change from Baseline to Week 12 | -0.9 (2.98) | -3.8 (8.66) | -1.5 (3.00) | -2.3 (5.40)
Statistical Analysis 1: Comparison: Placebo vs VAY736 Combined; Per protocol the primary analysis was between placebo and the combined VAY736 groups at Week 12; Test type: Superiority; p = 0.678, repeated measures Bayesian analysis; with baseline as a covariate; Mean Difference (Final Values) = -0.93, 95% CI 2-sided [-5.007 to 3.180], Standard Deviation 2.058

2. Secondary Outcome: Change in EULAR Sjögren's Syndrome Patient Response Index (ESSPRI)
Description: The ESSPRI is a patient self-reported outcome measure to assess dryness, limb pain, fatigue and mental fatigue, where each of the domains normally reported as 0 (not at all) to 10 (extremely severe). The final ESSPRI score is the average of three: dryness, pain and fatigue. A reduction from baseline indicates the improvement of symptoms. During the study all individual scores were reported as 1 to 10 instead. A linear transformation was reported to map the scores to the range of 0-10.
Time Frame: Baseline, week 12
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | VAY736 3 mg/kg | VAY736 10 mg/kg
Number analyzed (Participants) | 9 | 6 | 12
units on a scale
  Baseline | 5.967 (2.2179) | 6.049 (1.2759) | 6.235 (1.5379)
  Week 12 | 5.926 (1.5822) | 6.173 (1.4753) | 4.568 (2.5966)
  Change from Baseline to Week 12 | -0.041 (1.7805) | 0.123 (1.0120) | -1.667 (1.8918)

3. Secondary Outcome: Change in Short Form (36) Health Survey (SF-36)
Description: The SF-36 is a 36-item, patient self-reported outcome measure (questionnaires) of patient health. The outcome of the questionnaires in eight scales results in two summary scores, physical component and mental component, both ranging from 0 - 100. An increase from baseline in either component summary score indicates reduced disease burden.
Time Frame: Baseline, week 12
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | VAY736 3 mg/kg | VAY736 10 mg/kg
Number analyzed (Participants) | 9 | 6 | 12
units on a scale
  Physical component score: Baseline | 46.886 (6.3905) | 39.445 (4.2857) | 46.015 (9.3533)
  Physical component score: Week 12 | 44.788 (8.3513) | 45.493 (7.3060) | 47.671 (9.2804)
  Physical component score: Change from Baseline | -2.098 (7.9084) | 6.048 (4.7189) | 1.656 (5.4113)
  Mental component score: Baseline | 36.913 (15.2776) | 37.517 (6.8994) | 43.628 (11.3667)
  Mental component score: Week 12 | 41.012 (13.2991) | 40.170 (11.9815) | 46.700 (11.3182)
  Mental component score: Change from Baseline | 4.099 (5.3361) | 2.653 (17.1261) | 3.073 (11.5823)

4. Secondary Outcome: Change in Multidimensional Fatigue Inventory (MFI)
Description: The MFI is a patient self-reported outcome measure (questionnaires) to assess fatigue covering the following dimensions: General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Motivation and Reduced Activity. Each dimension has a posible range from 4-20. A reduction from baseline in MFI indicates improvement.
Time Frame: Baseline, week 12
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | VAY736 3 mg/kg | VAY736 10 mg/kg
Number analyzed (Participants) | 9 | 6 | 12
units on a scale
  General Fatigue: Baseline | 14.0 (4.72) | 17.0 (2.37) | 15.9 (3.34)
  General Fatigue: Week 12 | 12.8 (4.84) | 14.2 (6.40) | 12.4 (3.99)
  General Fatigue: Change from Baseline | -1.2 (1.64) | -2.8 (5.04) | -3.5 (4.12)
  Physical Fatigue: Baseline | 12.9 (4.14) | 15.7 (2.34) | 14.2 (3.41)
  Physical Fatigue: Week 12 | 12.2 (3.99) | 11.2 (5.15) | 10.4 (4.66)
  Physical Fatigue: Change from Baseline | -0.7 (1.32) | -4.5 (6.57) | -3.8 (4.77)
  Mental Fatigue: Baseline | 11.9 (4.78) | 14.3 (3.78) | 13.0 (3.28)
  Mental Fatigue: Week 12 | 11.7 (4.12) | 11.3 (4.18) | 9.8 (5.17)
  Mental Fatigue: Change from Baseline | -0.2 (2.95) | -3.0 (6.07) | -3.2 (5.84)
  Reduced motivation: Baseline | 12.4 (4.93) | 12.3 (3.93) | 10.9 (2.68)
  Reduced motivation: Week 12 | 12.0 (5.32) | 10.0 (4.52) | 9.8 (4.97)
  Reduced motivation: Change from Baseline | -0.4 (2.40) | -2.3 (4.50) | -1.1 (4.56)
  Reduced activity: Baseline | 11.8 (2.86) | 10.8 (1.72) | 12.2 (2.69)
  Reduced activity: Week 12 | 10.4 (3.81) | 8.7 (3.61) | 9.3 (5.08)
  Reduced activity: Change from Baseline | -1.3 (1.80) | -2.2 (4.83) | -2.9 (4.25)

5. Secondary Outcome: Change in the Physician's Global Assessment of Overall Disease Activity by Means of Visual Analog Scale (VAS)
Description: The visual analogue scale used is a 100 mm VAS ranging from "no disease" (0 mm) to "maximal disease activity" (100 mm).
Time Frame: Baseline, week 12
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | VAY736 3 mg/kg | VAY736 10 mg/kg
Number analyzed (Participants) | 9 | 6 | 12
units on a scale
  Baseline | 57.3 (17.73) | 66.2 (17.53) | 65.0 (11.74)
  Week 12 | 59.8 (23.35) | 43.0 (23.82) | 48.5 (17.33)
  Change from Baseline to Week 12 | 2.4 (12.21) | -23.2 (31.10) | -16.5 (18.96)

6. Secondary Outcome: Change in the Patient's Global Assessment of Overall Disease Activity by Means of Visual Analog Scale (VAS)
Description: The visual analogue scale used is a 100 mm VAS ranging from "no disease" (0 mm) to "maximal disease activity" (100 mm).
Time Frame: Baseline, week 12
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | VAY736 3 mg/kg | VAY736 10 mg/kg
Number analyzed (Participants) | 9 | 6 | 12
units on a scale
  Baseline | 56.2 (24.86) | 67.2 (13.69) | 59.8 (24.30)
  Week 12 | 55.2 (21.57) | 44.2 (22.75) | 40.8 (20.49)
  Change from Baseline to Week 12 | -1.0 (17.71) | -23.0 (25.73) | -19.0 (21.08)

7. Secondary Outcome: VAY736 Serum Concentration - AUCinf
Description: The area under the serum concentration-time curve from time zero to infinity [mass × time / volume]. The concentration of VAY736 was measured in the serum.
Time Frame: 0, 1, 2, 3, 6, 9, 12, 16, 20, 24 and approximately 52 weeks.
Population: PK analysis set
Measure: Median (Full Range); unit: day*ug/mL
Groups:
- Open Label VAY736: Open label VAY736 10mg/kg
Arm/Group | VAY736 3 mg/kg | VAY736 10 mg/kg | Open Label VAY736
Number analyzed (Participants) | 6 | 12 | 5
day*ug/mL | 389 [186 to 457] | 1140 [515 to 1610] | 971 [849 to 1340]

8. Secondary Outcome: VAY736 Serum Concentration - AUClast
Description: The area under the serum concentration-time curve from time zero to the time of the last quantifiable concentration [mass × time / volume]. The concentration of VAY736 was measured in the serum.
Time Frame: 0, 1, 2, 3, 6, 9, 12, 16, 20, 24 and approximately 52 weeks.
Population: PK analysis set
Measure: Median (Full Range); unit: day*ug/mL
Arm/Group | VAY736 3 mg/kg | VAY736 10 mg/kg | Open Label VAY736
Number analyzed (Participants) | 6 | 12 | 5
day*ug/mL | 385 [184 to 457] | 1140 [514 to 1610] | 971 [848 to 1340]

9. Secondary Outcome: VAY736 Serum Concentration - CL
Description: The systemic (or total body) clearance from serum following intravenous administration [volume / time]. The concentration of VAY736 was measured in the serum.
Time Frame: 0, 1, 2, 3, 6, 9, 12, 16, 20, 24 and approximately 52 weeks.
Population: PK analysis set
Measure: Median (Full Range); unit: L/day
Arm/Group | VAY736 3 mg/kg | VAY736 10 mg/kg | Open Label VAY736
Number analyzed (Participants) | 6 | 12 | 5
L/day | 0.594 [0.427 to 0.844] | 0.584 [0.550 to 1.30] | 0.686 [0.427 to 0.750]

10. Secondary Outcome: VAY736 Serum Concentration - Cmax
Description: The observed maximum serum concentration following drug administration [mass / volume]. The concentration of VAY736 was measured in the serum.
Time Frame: 0, 1, 2, 3, 6, 9, 12, 16, 20, 24 and approximately 52 weeks.
Population: PK analysis set
Measure: Median (Full Range); unit: ug/mL
Arm/Group | VAY736 3 mg/kg | VAY736 10 mg/kg | Open Label VAY736
Number analyzed (Participants) | 6 | 12 | 5
ug/mL | 65.0 [45.4 to 76.5] | 213 [150 to 283] | 205 [174 to 217]

11. Secondary Outcome: VAY736 Serum Concentration - T1/2
Description: Apparent terminal half-life, determined as the ln2/lambda_z or 0.693/lambda_z. The concentration of VAY736 was measured in the serum.
Time Frame: 0, 1, 2, 3, 6, 9, 12, 16, 20, 24 and approximately 52 weeks.
Population: PK analysis set
Measure: Median (Full Range); unit: days
Arm/Group | VAY736 3 mg/kg | VAY736 10 mg/kg | Open Label VAY736
Number analyzed (Participants) | 6 | 12 | 5
days | 8.43 [6.99 to 13.8] | 9.51 [5.38 to 15.2] | 11.0 [4.94 to 17.4]

12. Secondary Outcome: VAY736 Serum Concentration - Tmax
Description: The time to reach the maximum concentration after drug administration [time]. The concentration of VAY736 was measured in the serum.
Time Frame: 0, 1, 2, 3, 6, 9, 12, 16, 20, 24 and approximately 52 weeks.
Population: PK analysis set
Measure: Median (Full Range); unit: hours
Arm/Group | VAY736 3 mg/kg | VAY736 10 mg/kg | Open Label VAY736
Number analyzed (Participants) | 6 | 12 | 5
hours | 2.03 [2.00 to 2.20] | 2.03 [2.00 to 2.30] | 2.10 [2.02 to 2.17]

13. Secondary Outcome: VAY736 Serum Concentration - Vz
Description: The volume of distribution during the terminal elimination phase following intravenous administration [volume]. The concentration of VAY736 was measured in the serum.
Time Frame: 0, 1, 2, 3, 6, 9, 12, 16, 20, 24 and approximately 52 weeks.
Population: PK analysis set
Measure: Median (Full Range); unit: L
Arm/Group | VAY736 3 mg/kg | VAY736 10 mg/kg | Open Label VAY736
Number analyzed (Participants) | 6 | 12 | 5
L | 7.83 [6.55 to 10.7] | 8.68 [7.15 to 12.4] | 10.3 [4.93 to 18.6]

14. Primary Outcome: Overall Incidence of Adverse Events
Description: Number of subjects with Adverse Events during the double blind treatment period.
Time Frame: Baseline to Week 24
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | VAY736 3 mg/kg | VAY736 10 mg/kg | VAY736 Combined
Number analyzed (Participants) | 9 | 6 | 12 | 18
Participants
  Subjects with AEs | 8 | 6 | 11 | 17
  Subjects with AEs within 24hr of infusion | 2 | 6 | 11 | 17
  Subjects with AEs post 24hr of infusion | 8 | 6 | 8 | 14
  Subjects with Study drug-related AEs | 5 | 6 | 11 | 17
  Subjects with Infusion related AEs | 1 | 6 | 9 | 15

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date subject has provided informed consent until end of study (Week 28 or when B cell recovery was demonstrated, up to 3 years).
Description: All AEs were reported until week 52. After week 52 only AEs related to VAY736 and AEs related to infection, potential malignant events and neutropenia were recorded.
Groups:
- Placebo: Placebo
- VAY736 3mg/kg: VAY736 3mg/kg
- VAY736 10mg/kg: VAY736 10mg/kg
- Open Label VAY736 10mg/kg: Open label VAY736 10mg/kg
Arm/Group | Placebo | VAY736 3mg/kg | VAY736 10mg/kg | Open Label VAY736 10mg/kg
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6 | 0/12 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/9 | 2/6 | 0/12 | 1/5
Other Adverse Events (participants affected / at risk) | 9/9 | 6/6 | 11/12 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=9) | VAY736 3mg/kg (N=6) | VAY736 10mg/kg (N=12) | Open Label VAY736 10mg/kg (N=5)
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ovarian cyst torsion (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=9) | VAY736 3mg/kg (N=6) | VAY736 10mg/kg (N=12) | Open Label VAY736 10mg/kg (N=5)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Chalazion (Eye disorders) | 0 | 1 | 0 | 0
Keratitis (Eye disorders) | 0 | 1 | 0 | 0
Vitreous detachment (Eye disorders) | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Auriculotemporal syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Noninfective sialoadenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 5 | 4 | 5
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 1 | 1 | 0 | 0
Urogenital infection bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 6 | 9 | 3
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 2 | 2 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-10-31): https://cdn.clinicaltrials.gov/large-docs/20/NCT02149420/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-11): https://cdn.clinicaltrials.gov/large-docs/20/NCT02149420/SAP_001.pdf